CLINICAL TRIAL: NCT01915264
Title: Glucobay M - Evaluation of Safety and Effectiveness in Type 2 Diabetes Not Well Controlled on Monotherapy in Real Life Practice
Acronym: GLORY
Status: Withdrawn | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16445; GB1310IN (Other: company intermal)
Record Dates: First submitted 2013-07-25; First posted 2013-08-02 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus; Type 2 Diabetes; Acarbose (25/50mg) and Metformin (500mg) in fixed dose combination
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Acarbose; Metformin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Acarbose/Metformin (Glucobay M, BAY81-9783)

INTERVENTIONS:
Drug: Acarbose/Metformin (Glucobay M, BAY81-9783) — Acarbose (25/50mg) and Metformin (500mg) in fixed dose combination.

SUMMARY:
The study is designed as non interventional to collect data on the safety especially, severe hypoglycemia or documented symptomatic hypoglycemic episodes and effectiveness of acarbose/metformin fixed-dose combination under real-life treatment condition in large sample of type-2 diabetes patients in India. The study objective is to evaluate severe hypoglycemia or documented symptomatic or asymptomatic hypoglycemic events reported as adverse events. The study will begin after the study approval by ethics committee. All patients with type 2 diabetes on acarbose or metformin monotherapy and prescribed Glucobay M will be included in study after taking the informed consent. Patients will be observed for up to 24 weeks (2 weeks).The study involves general examination of patients, collection of data like history of disease, concomitant medication, drug dose etc. The study is planned to enroll 10000 subjects from multiple study centers spread across India. The study data will be analyzed with appropriate statistical methods.

ELIGIBILITY:
Inclusion Criteria:

* Patient will be enrolled after the decision to administer acarbose/metformin fixed dose combination for type-2 diabetes management has been made by the attending physician on the basis of best clinical practice and patient needs.
* Willing to give informed consent for participating in this study

Exclusion Criteria:

* Patients receiving anti-diabetic medication other than acarbose, or metformin monotherapy at the time of enrollment in the study will be excluded. However, during observation period, any additional anti-diabetics medication administered by the attending physician will be allowed & recorded in case record form.
* Patient receiving acarbose/metformin fixed dose combination during 3-months prior to enrollment.
* Exclusion criteria should be read in conjunction with local product information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of severe hypoglycemia or documented symptomatic or asymptomatic hypoglycemic events reported as adverse events | 24 weeks

SECONDARY OUTCOMES:
Incidence of adverse events other than hypoglycemia reported | 24 weeks
Mean change in HbA1c level | baseline and 24 weeks
Mean change in fasting blood sugar | baseline and 24 weeks
Mean change in postprandial blood sugar | baseline and 24 weeks
Mean change in body weight | baseline and 24 weeks
Mean change in serum LDL(low-density lipoprotein) cholesterol | baseline and 24 weeks
Mean change in serum triglyceride | baseline and 24 weeks
Mean change in serum HDL (High density lipoproteins) cholesterol | baseline and 24 weeks
Change in percent satisfaction to the therapy from baseline as measured by 5 point satisfaction scale | baseline and 24 weeks
Number of patient with adverse event (Tolerability) | Baseline and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer